CLINICAL TRIAL: NCT06125275
Title: Pattern of Acute Antipsychotic Drug- Toxicity in Children at Assiut University Children Hospital
Brief Title: Pattern of Acute Antipsychotic Drug- Toxicity in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ramadan Hussein Mohamed, 71515,Assiut, Assiut University
Other Study IDs: Antipsychotic Drug- Toxicity
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Antipsychotic Drug- Toxicity
Keywords: Antipsychotic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pattern of Acute Antipsychotic Drug- Toxicity in Children at Assiut University Children Hospital.

* Determine the pattern and outcome of acute antipsychotic drug- toxicity of children who are admitted to The emergency department of Assiut University Children Hospital (AUCH).
* Estimate prevalence of acute antipsychotics drug-toxicity in children and adolescents at AUCH.

DETAILED DESCRIPTION:
Acute poisoning in pediatrics is very common as it is one of the prominent causes of mortality and morbidity worldwide as, children are curious and they explore at home and around. Acute poisoning has also been the 3rd most common treated injury for children less than 16 years in the emergency units. Accidental ingestion is one of the most important causes of poisoning in children and is most prevalent between 1-5 year olds. During adolescence, medications used for committing suicide are the main cause of poisoning.

Drug ingestion is the commonest cause of acute poisoning among children according to poison control centers records all over the world. A great percent of hospital admission cases involves drug poisoning, particularly with psychotropic drugs such as sedatives, antidepressants, and neuroleptics.

Antipsychotics are primary used to treat agitated behavior , various neurological conditions (motor tics ,chorea and dystonia),schizophrenia, manic phase of bipolar disorders; however they are often used to treat nausea, vomiting and headache. Antipsychotics toxic effects include anticholinergic and extrapyramidal syndromes as well as CNS and cardiovascular depression.

Antipsychotics are classified as ""typical"" or ""atypical."" They are also classified by their chemical structure as first-generation, including butyrophenones (droperidol, haloperidol) and phenothiazines (chlorpromazine, promethazine), and second generation such as olanzapine, risperidone, quetiapine, and more recently ziprasidone and aripiprazole.

Second-generation antipsychotics, or ''atypical antipsychotics,'' were introduced in 1989 and were anticipated to be equally effective for treatment of psychosis.They also had the advertised advantage of fewer extrapyramidal side effects such as dystonias, akathisia, parkinsonism, and tardive dyskinesia, at therapeutic dosing.

These medications are now first-line therapy in the treatment of schizophrenia and are additionally being used in a wide array of conditions in both adults and children, including bipolar disorder, tic disorders, eating disorders, obsessive-compulsive disorder, and developmental disorders such as autism. Risperidone and aripiprazole were approved by the FDA in 2006 and 2009, respectively, to treat irritability associated with Autism spectrum disorder (ASD).

Antipsychotics overdose is common in Western society. In 2010, poison control centers in the US received about 43 000 calls complaining of atypical antipsychotics overdose. The actual incidence of atypical antipsychotics overdose is greater than announced, due to underreporting. Overdose of an atypical antipsychotic is presented clinically with multiple disorders as CNS depression, tachycardia and orthostatic hypotension.

Supportive measures as maintaining patent airway, assessment of breathing, maintaining adequate circulation are necessary before confirmation of intoxication. Evaluation and management of antipsychotic drugs toxicities needs high level of suspicion, careful history taking, proper examination, and investigations to improve the outcome of such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of exposure to antipsychotic drugs aged from 1month to 18 years old, who presented to emergency department.
2. Both sexes.
3. Diagnosis is according to clinical features suggestive of possible antipsychotic drug- toxicity.

Exclusion Criteria:

1. neonates less than one month .
2. History of chronic exposure.
3. Food poisoning and other poisonous.
4. Other drugs toxicity.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: atients with history of exposure to antipsychotic drugs aged from 1month to 18 years old, who presented to emergency department
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Determine the pattern and outcome of acute antipsychotic drug- toxicity of children who are admitted to The emergency department of Assiut University Children Hospital (AUCH). | Baseline
  Estimate prevalence of acute antipsychotics drug-toxicity in children and adolescents at AUCH

REFERENCES:
- [Background] Berta GN, Di Scipio F, Bosetti FM, Mognetti B, Romano F, Carere ME, Del Giudice AC, Castagno E, Bondone C, Urbino AF. Childhood acute poisoning in the Italian North-West area: a six-year retrospective study. Ital J Pediatr. 2020 Jun 11;46(1):83. doi: 10.1186/s13052-020-00845-0. PMID 32527281
- [Background] Gummin DD, Mowry JB, Spyker DA, Brooks DE, Fraser MO, Banner W. 2016 Annual Report of the American Association of Poison Control Centers' National Poison Data System (NPDS): 34th Annual Report. Clin Toxicol (Phila). 2017 Dec;55(10):1072-1252. doi: 10.1080/15563650.2017.1388087. Epub 2017 Nov 29. PMID 29185815
- [Background] Evoy KE, Peckham AM, Covvey JR, Tidgewell KJ. Gabapentinoid Pharmacology in the Context of Emerging Misuse Liability. J Clin Pharmacol. 2021 Aug;61 Suppl 2:S89-S99. doi: 10.1002/jcph.1833. PMID 34396549